CLINICAL TRIAL: NCT03632317
Title: A Phase 2 Study of Panobinostat in Combination With Everolimus for Children and Young Adults With Gliomas Harboring H3.3 or H3.1 K27M Mutation
Brief Title: A Study of Panobinostat in Combination With Everolimus for Children and Young Adults With Gliomas
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2018.006; HUM00140679 (Other: University of Michigan)
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Glioma; Diffuse Intrinsic Pontine Glioma
Keywords: H3.1K27M; H3.3K27M; diffuse intrinsic pontine glioma; DIPG; high-grade glioma; pediatric glioma; H3K27M; panobinostat
MeSH Terms: conditions — Glioma; Diffuse Intrinsic Pontine Glioma | interventions — Panobinostat; Everolimus

STUDY DESIGN:
Intervention Model Description: Patients will be divided into two stratums; newly diagnosed high-grade glioma or DIPG after radiation (stratum A) and recurrent/progressive glioma (grade II-IV, including DIPG) (stratum B).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Panobinostat and Everolimus (Experimental): Panobinostat daily M, W, F for 2 weeks every 28 days for the first cycle (28 days). After first cycle Panobinostat daily M, W, F for 2 weeks every 28 days combined with Everolimus daily.
  Interventions: Drug: Panobinostat; Drug: Everolimus

INTERVENTIONS:
Drug: Panobinostat — 30 mg/m^2
Drug: Everolimus — 3.0 mg/m^2

SUMMARY:
This phase 2 trial will evaluate the activity of Panobinostat in combination with Everolimus for children with gliomas harboring H3.1 or H3.3K27M mutation, including newly diagnosed high-grade glioma or DIPG (diffuse intrinsic pontine glioma) after radiation (stratum A) and recurrent/progressive glioma (grade II-IV, including DIPG) (stratum B).

ELIGIBILITY:
Inclusion Criteria:

* All patients and/or a legal guardian must sign institutionally approved written informed consent and assent documents.
* Patient must be greater than 2 years and less than 30 years
* BSA (body surface area) greater than 0.3 m2
* Functional status: Karnofsky > 50% for patients > 16 years of age and Lansky > 50% for patients < 16 years of age (Karnofsky and Lansky is a scoring system used to quantify the general well being of cancer patients where 100% represents perfect health and 0% represents death). Neurologic deficits in patients with CNS tumors must have been relatively stable for a minimum of 7 days. Patients who are unable to walk because of paralysis, but who are able to sit in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
* Adequate bone marrow function
* Adequate liver function
* Adequate renal and metabolic function
* Urine protein:creatinine (UPC) ratio of < 1; or a urinalysis that is negative for protein; or 24-hour urine protein level < 1000 mg/dL
* Patients must have Magnesium > 1.5 mg/dL and potassium > 3.5 mmol/L
* Patients with known seizure disorder must have seizures adequately controlled with non- enzyme inducing antiepileptic medications
* No increase in steroid dose within the past 7 days.
* STRATUM A: histological confirmation of a newly diagnosed high-grade glioma or DIPG or STRATUM B: histological confirmation of a recurrent or progressive grade II-IV glioma (including DIPG) [histology can come from tissue at diagnosis or relapse]
* Primary brain or spine tumor are eligible, including tumors with metastases, multiple lesions
* Patients must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy.
* Myelosuppressive chemotherapy: Must not have received within 3 weeks (6 weeks if prior nitrosourea).
* Hematopoietic growth factors: At least 7 days since the completion of therapy with a growth factor, 14 days for long-acting (e.g. PEG-filgrastim)
* Biologic (anti-neoplastic agent): At least 7 days or 3 half-lives (whichever is longer) since the completion of therapy with a biologic agent.
* Radiation therapy: Strata A: ≥ 2 weeks and ≤ to 12 weeks must have elapsed from radiation. Strata B: ≥ 2 weeks must have elapsed from focal radiation.
* Surgery: > 3 weeks from major surgery. If recent craniotomy, adequate wound healing must be determined by neurosurgical team.
* Autologous Stem Cell Transplant or Rescue: No evidence of active graft vs. host disease and ≥ 4 weeks must have elapsed.
* H3K27M mutation: Participants must have a mutation in H3.3 K27M or H3.1 K27M as identified by tumor (FFPE or fresh, diagnosis or relapse tissue, but relapse tissue preferred) sequencing, or by CLIA-certified immunohistochemistry staining positive for H3K27M, as defined by review by U of M neuro-pathology.

Exclusion Criteria:

* Patients who are breastfeeding, pregnant or refuse to use an effective form of birth control are excluded. Abstinence is considered an effective form of birth control.
* Patients with uncontrolled infection are excluded.
* Inability to swallow oral pill (panobinostat does not have liquid formulation).
* Other medications: Patients receiving other anti-neoplastic agents are excluded; patients on enzyme-inducing anticonvulsive agents are excluded; patients requiring strong CYP3A4 or PGP inducers or inhibitors are excluded; patients on steroids for symptom management must be on a stable dose for 7 days prior to start of treatment.
* Allogeneic stem cell transplant: Patients within 1 year of allogeneic stem cell transplant, patients with active GVHD or requiring immunosuppression are excluded.
* Previous hypersensitivity to rapamycin or rapamycin derivatives.
* Baseline QTc of >450 msec on EKG OR electrolyte imbalance predisposing to QTc prolongation (baseline ≥ Grade 1 hypokalemia or hyperkalemia; and baseline ≥ Grade 2 Ca++, Mg++, phosphate abnormalities). Repletion/correction is allowed to achieve eligibility. Use of QTC prolonging medications will be monitored throughout the trial.

Ages: 2 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Median Progression Free Survival (PFS) at 1 Year | 1year
  Median PFS at 1 year for stratum A will be measured. Progression is defined as > 25% increase in the size of the tumor or appearance of new lesions.
Median Progression Free Survival (PFS) at 2 Years | 2years
  Median PFS at 1 year for stratum A will be measured. Progression is defined as > 25% increase in the size of the tumor or appearance of new lesions.
Overall Survival at 1Year | 1year
  The proportion of patients alive at 1 year for stratum A.
Overall Survival at 2Years | 2years
  The proportion of patients alive at 2 years for stratum A.
Overall Response Rate (ORR) After Two Cycles of Panobinostat + Everolimus | 84 Days
  Overall Response Rate (ORR) After Two Cycles of Panobinostat + Everolimus for stratum B. Overall response is defined as a partial or complete response. Partial response is defined as a ≥50% decrease in size of tumor in comparison to baseline measurements. Complete response is defined as the disappearance of all abnormal signal. This includes return to normal size of the brainstem for brainstem lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Carl Koschmann, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No